CLINICAL TRIAL: NCT02916251
Title: Randomised, Sequential, Cross-over Trial Assessing PK and PD Responses After Micro-doses of ZP4207 Administered s.c. to Patients With T1D Under eu- and Hypoglycemic Conditions and With Reference to Freshly Reconstituted Lyophilized Glucagon
Brief Title: ZP4207(Dasiglucagon) Administered to T1D Patients to Assess the PK and PD Compared to Marketed Glucagon
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ZP4207-16098
Record Dates: First submitted 2016-09-08; First posted 2016-09-27 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Mellitus Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — dasiglucagon; Glucagon

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ZP4207(dasiglucagon) (Experimental): Intervention: ZP4207(dasiglucagon) glucagon analogue (4 mg/mL) planned doses: 0.03, 0.08, 0.2 and 0.6 mg at euglycemic and hypoglycemic conditions.
  Interventions: Drug: ZP4207(dasiglucagon) glucagon analogue
- Glucagon (Native glucagon) (Active Comparator): Intervention: Glucagon (Native glucagon) 1 mg/mL as active comparator planned doses: 0.03, 0.08 and 0.2 mg at euglycemic conditions.
  Interventions: Drug: Glucagon (Native glucagon)

INTERVENTIONS:
Drug: ZP4207(dasiglucagon) glucagon analogue — Cross-over design with single s.c. administration in euglycemic and hypoglycemic T1D
  Other Names: dasiglucagon
  Arms: ZP4207(dasiglucagon)
Drug: Glucagon (Native glucagon) — Cross-over design with single s.c. administration in euglycemic T1D
  Other Names: Lilly Glucagon
  Arms: Glucagon (Native glucagon)

SUMMARY:
The trial is a single-centre, randomised, sequential, cross-over trial assessing pharmacokinetic and pharmacodynamic responses after micro-doses of ZP4207 (dasiglucagon*) administered subcutaneously to patients with type 1 diabetes mellitus under euglycaemic and hypoglycaemic conditions and compared to marketed glucagon.

*dasiglucagon is the proposed International Nonproprietary Name (pINN) for ZP4207

DETAILED DESCRIPTION:
Seventeen (17) adult patients with T1DM treated with continuous subcutaneous insulin infusion (insulin pumps, CSII) will be randomized and take part at four dosing visits. The dosing visits are separated by 3-7 days. For the three lowest dose levels (0.03 mg, 0.08 mg, and 0.2 mg) the patients will receive two doses of ZP4207(dasiglucagon) (the first at euglycaemic and the second at hypoglycaemic conditions) and one dose of glucagon at euglycaemic conditions at visit 2-4. The first two dose administrations (Day 1, visit 2-4) will be separated by at least five hours. The third dose, which is ZP4207(dasiglucagon) during hypoglycemia, will for all dosing visits be administered the next morning after a standardized carbohydrate-rich meal in the evening before. The patients will stay at the clinical site over night between Day 1 and Day 2. The dose of 0.6 mg will only be administered for ZP4207(dasiglucagon). The order of the micro-dose levels as well as the order of the treatment, ZP4207(dasiglucagon) vs. glucagon, will be randomized. For all patients the 0.6 mg dose of ZP4207(dasiglucagon) will be administered at visit 5.

For each dose level there will be 2 sets of PK/PD profiles for ZP4207(dasiglucagon), one initiated during euglycaemia and another during hypoglycaemia. Each patient enrolled will therefore provide a total of 11 PK/PD profiles covering four different dose levels; 8 profiles from ZP4207(dasiglucagon) and 3 profiles from glucagon

ELIGIBILITY:
Inclusion Criteria:

To be included in the trial, patients have to fulfil all of the following criteria:

1. Signed and dated informed consent obtained before any trial-related activities. (Trial-related activities are any procedures that would not have been performed during normal management of the patient).
2. Male and female patients with T1DM for at least 1 year, as defined by the American Diabetes Association1.
3. Age between 18 and 64 years, both inclusive.
4. HbA1c < 8.5%.
5. C-peptide negative defined as below the lower limit of quantification.
6. Stable insulin regimen via an insulin infusion pump for at least 1 month prior to screening.
7. Weight between 60 kg and 90 kg, both inclusive.
8. Patients in good health according to age (medical history, physical examination, vital signs, 12-lead ECGs, lab assessments), as judged by the Investigator.-

Exclusion Criteria:

Patients meeting any of the following criteria during screening evaluations will be excluded from trial participation:

1. Unable to provide informed consent (e.g., impaired cognition or judgement).
2. Patients with mental incapacity or language barriers which preclude adequate understanding or cooperation, who are unwilling to participate in the trial, or who in the opinion of the Investigator should not participate in the trial.
3. Receipt of any medicinal product in clinical development within 3 months prior screening.
4. Previous exposure to ZP4207(dasiglucagon) or previously randomized to this trial.
5. Known or suspected allergy to trial product(s) or related products.
6. History of adverse reaction to glucagon (including allergy) besides nausea and vomiting.
7. History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction.
8. New onset clinically significant illness within 4 weeks prior to screening, as judged by the Investigator.
9. History of liver disease that is expected to interfere with the anti-hypoglycemia action of glucagon (e.g., liver failure or cirrhosis). Other liver disease (i.e., active hepatitis, steatosis, active biliary disease, any tumor of the liver, hemochromatosis, glycogen storage disease) may exclude the patient if it causes significant compromise to liver function or may do so in an unpredictable fashion.
10. Any history or presence of clinically relevant cardiovascular, pulmonary, respiratory, gastrointestinal, renal, metabolic, endocrinological (with the exception of conditions associated with diabetes mellitus), haematological, dermatological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynaecologic (if female), or infectious disease, or signs of acute illness as judged by the Investigator.
11. Clinically significant abnormal haematology, biochemistry or urinalysis screening tests, as judged by the Investigator. In particular, elevated liver enzymes (AST or ALT > 2 times the upper limit of normal, or bilirubin >1.5 the upper limit of normal) or impaired renal function (elevated serum creatinine values above the upper limit of normal).
12. Hypertension with systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg (excluding white-coat hypertension; therefore, if a repeated measurement shows values within the range, the patient can be included in the trial); a heart rate at rest outside the range of 50-90 beats per minute.
13. Clinically significant abnormal standard 12-lead electrocardiogram (ECG) after 5 minutes resting in supine position at screening, as judged by the Investigator.
14. Proliferative retinopathy or maculopathy and/or severe neuropathy, in particular autonomic neuropathy, as judged by the Investigator.
15. Inadequate venous access as determined by trial nurse or physician at time of screening
16. Any factors that, in the judgment of the Principal Investigator, would interfere with trial endpoints or the safe completion of the trial procedures.
17. Severe hypoglycaemic events within one year prior to screening, as judged by the Investigator.
18. Increased risk of thrombosis, e.g. patients with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator.
19. Significant history of alcoholism or drug abuse as judged by the Investigator or consuming more than 24 g alcohol per day for men, or more than 12 g alcohol per day for women.
20. A positive result in the alcohol and/or urine drug screen at the screening visit.
21. Habitual smoking, i.e., daily smoking or more than 7 cigarettes/week within the last 3 months prior to screening. Patients have to accept refraining from smoking while at the clinical site.
22. History of cystic fibrosis, pancreatitis, pancreatic tumor, or any other pancreatic disease besides T1DM
23. History of pheochromocytoma.
24. History of adrenal disease or tumor.
25. Positive to the screening test for Hepatitis Bs antigen or Hepatitis C antibodies and/or a positive result to the test for HIV-1/2 antibodies or HIV-1 antigen.
26. The use of any non-prescribed systemic or topical medication, except routine vitamins and occasional use of acetylsalicylic acid and paracetamol within 2 weeks prior to randomization (and if female with the exception of hormonal contraception or menopausal hormone replacement therapy).
27. Donation of blood or plasma in the past month, or in excess of 500 mL within 12 weeks prior to screening.
28. Male who is sexually active and not surgically sterilized who or whose partner(s) is not using highly effective contraceptive methods (highly effective contraceptive measures include surgical sterilisation, hormonal intrauterine devices [coil], oral hormonal contraceptives, each in combination with spermicide-coated condoms), or who is not willing to refrain from sexual intercourse from the first dosing until the end of the trial (Visit 6).
29. Females of childbearing potential who are pregnant (positive urine human chorionic gonadotropin [HCG]), breast-feeding or intend to become pregnant or are not using highly effective contraceptive methods (highly effective contraceptive methods are considered those with a failure rate less than 1% undesired pregnancies per year including surgical sterilisation, hormonal intrauterine devices (coil), oral hormonal contraceptives, sexual abstinence or a surgically sterilised partner). Females who are postmenopausal can participate in the study without using adequate contraceptive methods. Postmenopausal is defined as women aged < 52 years and being amenorrheic for more than one year with serum FSH level > 40 IU/L or aged >= 52 years and being amenorrheic for less than one year and with serum FSH level > 40 IU/L or aged >= 52 years being amenorrheic for more than one year.

    -

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-05 (Actual)

PRIMARY OUTCOMES:
PK endpoint for ZP4207(dasiglucagon) and baseline adjusted glucagon: AUC 0-240 min | AUC 0-240 min during all treatment periods (V2-V5)
  Area under the curve from 0-240 min
PK endpoint for ZP4207(dasiglucagon) and baseline adjusted glucagon: Cmax | Pre-dose, 5, 15, 30, 60, 90, 150 and 240 minutes post dosing. Peak of plasma concentration during all treatment periods (V2-V 5)
  max. concentration
PK endpoint for ZP4207(dasiglucagon) and baseline adjusted glucagon: tmax | Pre-dose, 5, 15, 30, 60, 90, 150 and 240 minutes post dosing. Time to peak plasma concentration during all treatment periods (V2-V5)
  Time to peak plasma concentration
PD endpoint: Plasma glucose profiles above baseline: AUE 0-240 min | Pre-dose, 10, 30, 50, 70, 90, 150, 240 minutes post dosing. AUE 0-240 min during all treatment periods (V2-V5)
  Area under the effect curve from 0-240 min
PD endpoint: Plasma glucose profiles above baseline: CEmax | Pre-dose, 10, 30, 50, 70, 90, 150, 240 minutes post dosing. Peak of plasma glucose concentration during all treatment periods (V2-V5)
  Max concentration effect
PD endpoint: Plasma glucose profiles above baseline: tmax | Pre-dose, 10, 30, 50, 70, 90, 150, 240 minutes post dosing Time to plasma glucose concentration during all treatment periods (V2-V5)
  Time to peak plasma glucose concentration

SECONDARY OUTCOMES:
PK endpoints for ZP4207(dasiglucagon) and baseline adjusted glucagon: MRT | Pre-dose, 5, 15, 30, 60, 90, 150 and 240 minutes post dosing. Mean residence time for ZP4207(dasiglucagon) and baseline adjusted glucagon during all treatment periods (V2-V5)
  Mean residence time
PK endpoints for ZP4207(dasiglucagon) and baseline adjusted glucagon: Vz/f, | Pre-dose, 5, 15, 30, 60, 90, 150 and 240 minutes post dosing. Volume of distribution of plasma ZP4207(dasiglucagon) or glucagon during all treatment periods (V2-V5)
  Volume of distribution
PK endpoints for ZP4207(dasiglucagon) and baseline adjusted glucagon: λz | Pre-dose, 5, 15, 30, 60, 90, 150 and 240 minutes post dosing. Terminal elimination rate constant of ZP4207(dasiglucagon) and baseline adjusted glucagon during all treatment periods (V2-V5)
  Terminal elimination rate constant
PK endpoints for ZP4207(dasiglucagon) and baseline adjusted glucagon: t½, | Pre-dose, 5, 15, 30, 60, 90, 150 and 240 minutes post dosing. Terminal plasma elimination half-life of ZP4207(dasiglucagon) or glucagon during all treatment periods (V2-V5)
  Terminal plasma elimination half-life
PK endpoints for ZP4207(dasiglucagon) and baseline adjusted glucagon: CL/f | Pre-dose, 5, 15, 30, 60, 90, 150 and 240 minutes post dosing. Total body clearance of plasma ZP4207(dasiglucagon) or glucagon during all treatment periods (V2-V5)
  Total body clearance
PK endpoints for ZP4207(dasiglucagon) and baseline adjusted glucagon: AUC 0-30min | AUC 0-30 min during all treatment periods (V2-V 5)
  Area under the curve from 0-30 min
PK endpoints for ZP4207(dasiglucagon) and baseline adjusted glucagon: AUC 0-inf | Pre-dose, 5, 15, 30, 60, 90, 150 and 240 minutes post dosing. AUC 0-inf during all treatment periods (V2-V 5)
  Area under the curve from 0-inf
Insulin concentrations before and after dosing with ZP4207(dasiglucagon) or glucagon: | Pre-dose, 5, 15, 30, 60, 90, 150 and 240 minutes post dosing. Insulin concentrations during all treatment periods (V2-V 5)
  Insulin concentrations
PD endpoints for ZP4207(dasiglucagon) and baseline adjusted glucagon: AUE 0-30min | AUE 0-240 min during all treatment periods (V2-V5)
  Area under the effect curve from 0-30 min
PD endpoints for ZP4207(dasiglucagon) and baseline adjusted glucagon: CE 30min | Concentration effect at 30 min during all treatment periods (V2-V5)
  Concentration effect at 30 min
PD endpoints for ZP4207(dasiglucagon) and baseline adjusted glucagon: t50%CE, early | Pre-dose, 10, 30, 50, 70, 90, 150, 240 minutes post dosing. Time to half concentration effect (t50%CE, early) during all treatment periods (V2-V5)
  Time to half concentration effect
PD endpoints for ZP4207(dasiglucagon) and baseline adjusted glucagon: t10%CE, late | Pre-dose, 10, 30, 50, 70, 90, 150, 240 minutes post dosing. Time to 90% decrease from peak concentration effect during all treatment periods (V2-V5)
  Time to 90% decrease from CEmax
PD endpoints: Percentage of patients achieving a plasma glucose increase of ≥20 mg/dL within 30 minutes after treatment | During all treatment periods (V2-V5) within 30 min after dosing
PD endpoints: Time to plasma glucose increase of ≥20 mg/dL | Pre-dose, 10, 30, 50, 70, 90, 150, 240 minutes post dosing. During all treatment periods (V2-V5) - time plasma glucose increase of ≥20 mg/dL after dosing
PD endpoints: Percentage of patients achieving a plasma glucose concentration ≥70 mg/dL within 30 minutes after treatment (insulin-induced hypoglycemia) | During all treatment periods (V2-V5) within 30 min after dosing (insulin-induced hypoglycemia)
PD endpoints: Time to plasma glucose concentration of ≥70 mg/dL (insulin-induced hypoglycemia) | Pre-dose, 10, 30, 50, 70, 90, 150, 240 minutes post dosing. During all treatment periods (V2-V5) - time plasma glucose increase of ≥70 mg/dL after dosing (insulin-induced hypoglycemia)
Safety endpoints: Number of participants with adverse events | Through study completion. The total trial duration for a patient will be about 5.5 to 12 weeks.
  Includes events from the first trial related activity after the patient has signed the informed consent until Follow up visit.
Safety endpoints: Local tolerability of injection site | Local tolerability assessed pre-dose (within 30 min) and at 0.5, 2, and 4 hours post-dose (each treatment visit and at Follow up visit).
  Findings in local tolerability by means of the following assessments:
  spontaneous pain
  * pain on palpation
  * itching
  * redness
  * oedema
  * induration/infiltration
  * other these assessments will be reported on a scale of 0 (none), 1 (mild), 2 (moderate) and 3 (severe)
Safety endpoints: Laboratory safety parameters | Through study completion. The total trial duration for a patient will be about 5.5 to 12 weeks.
  Haematology, biochemistry and urinalysis: Changes or findings from baseline (normal ranges) in clinical safety laboratory parameters during the study duration (from Screening, at treatment visits and at Follow up visit).
Safety endpoints: Physical examination | Through study completion. The total trial duration for a patient will be about 5.5 to 12 weeks.
  Physical examination: Changes or findings from baseline (normal ranges) in physical examination during the study duration (at Screening and Follow up visit).
  An examination of the following body systems will be performed:
  Head, ears, eyes, nose, throat (HEENT), incl thyroid gland Heart, lung, chest Abdomen Skin and mucosae Musculoskeletal system Nervous system Lymph node Other findings
Safety endpoints: Vital signs | Through study completion. The total trial duration for a patient will be about 5.5 to 12 weeks.
  Diastolic and systolic blood pressure (mmHg) are measured after at least 5 min rest in a supine position. At the screening visit blood pressure is measured in both arms. The blood pressure from the arm with the higher systolic value is transcribed into the CRF and this arm is used for all subsequent measurements of the patient's blood pressure in this trial.
  Pulse (beats per min) measured after at least 5 min rest in a supine position. Body temperature, tympanic (in Celsius). Respiratory frequency (RF/min). Changes or findings from baseline (normal ranges) in vital signs during the study duration (at Screening, at each treatment visit and at Follow up).
Safety endpoints: ECGs | Through study completion. The total trial duration for a patient will be about 5.5 to 12 weeks.
  A standard 12-lead electrocardiogram (ECG) will be performed. ECG parameters (Heart rate, PQ, QRS, QT, QTcB) and any abnormality will be recorded and described in the CRF including the Investigator's assessment of clinical significance ('abnormal, not clinically significant' or 'abnormal, clinically significant'). Clinically significant findings at the screening visit should be recorded as concomitant illness.
  At subsequent visits, any clinically significant deterioration of a pre-existing condition as well as any new clinically significant findings will be recorded as AEs.
  Changes or findings from baseline (normal ranges) (Screening visit and at Follow up) in ECGs during the study duration.
Safety endpoints: Antidrug antibodies incidences | Through study completion. The total trial duration for a patient will be about 5.5 to 12 weeks.
  Antidrug antibodies analyses will be performed. Changes or findings from baseline (normal ranges) in Antidrug antibodies incidences during the study duration (before first dosing, at last treatment visit and at Follow up).

CONTACTS AND LOCATIONS:
Overall Officials: Hövelmann Ulrike, MD, Principal Investigator — Profil Neuss GmbH Neuss, Germany, 41460
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided